CLINICAL TRIAL: NCT07160608
Title: Phase 2, Randomized, Double-Blind, Placebo-controlled, Parallel-Group, Multicenter Study to Evaluate the Safety and Efficacy of Tarperprumig in Adult Participants With Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis (I TRANSCEND)
Brief Title: Safety and Efficacy of Tarperprumig in Adult Participants With Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6722C00001; 2025-521706-17-00 (Other: EU CT); ALXN1820-ANCA-201 (Other: Alexion)
Record Dates: First submitted 2025-07-21; First posted 2025-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: ANCA-associated vasculitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis; IMP (Tarperprumig)
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tarperprumig Group 1 (Experimental): Participants will be administered tarperprumig dose regimen #1 or dose regimen #2.
  Interventions: Drug: Tarperprumig
- Tarperprumig Group 2 (Experimental): Participants will be administered tarperprumig dose regimen #1 or dose regimen #2.
  Interventions: Drug: Placebo; Drug: Tarperprumig
- Placebo Group 3 (Experimental): Participants will be administered placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo.
  Arms: Placebo Group 3; Tarperprumig Group 2
Drug: Tarperprumig — Participants will receive tarperprumig.
  Other Names: ALXN1820
  Arms: Tarperprumig Group 1; Tarperprumig Group 2

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of tarperprumig in participants with newly diagnosed or relapsing anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsing ANCA-associated vasculitis, GPA and MPA subtypes consistent with the 2022 ACR/EULAR classification criteria for GPA and MPA for whom treatment with rituximab or cyclophosphamide is considered.
* Positive test for antibodies to either PR3-ANCA or MPO-ANCA at Screening or in the past by a quantitative assay (for example, ELISA, bead assay).
* At least one major item, or at least 3 minor items, or at least 2 renal items in the BVAS.

Exclusion Criteria:

* Other systemic diseases that, in the judgment of the Investigator, constitute the primary illness, including but not limited to: eosinophilic granulomatosis with polyangiitis (EGPA), systemic lupus erythematosus, IgA nephropathy and/or IgA associated vasculitis with or without Henoch-Schonlein purpura, rheumatoid vasculitis, Sjogren's syndrome, anti-GBM disease, cryoglobulinemic vasculitis, autoimmune hemolytic anemia, or mixed connective tissue disease.
* Alveolar hemorrhage requiring invasive pulmonary ventilation support at Screening.
* Any diseases or conditions that, in the judgment of the Investigator, present a substantial clinical risk to participate in this study.
* For patients with a previous diagnosis of CKD, patients known to have a stable eGFR for greater than 3 months prior to Screening and a decline less than 25% of previous eGFR at Screening will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-10-06 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline through Week 70

SECONDARY OUTCOMES:
Number of Participants Achieving Disease Remission at Week 26 | Week 26
Number of Participants Achieving Sustained Remission at Week 52 | Week 52
Number of Participants Achieving a Birmingham Vasculitis Activity Score (BVAS) of 0 | Baseline through Week 52
Number of Participants Experiencing a Relapse After Previously Achieving Disease Remission at Week 26 | Week 26 through Week 70
Time to First Relapse After Having Achieved Disease Remission at Week 26 | Week 26 through Week 70
Change from Baseline in Vasculitis Damage Index | Baseline, Weeks 26, and 52
Time to First Occurrence of BVAS of 0 | Baseline through Week 52
Change from Baseline in BVAS | Baseline, Weeks 26, and 52
Change from Baseline in Estimated Glomerular Filtration Rate | Baseline, Weeks 26, and 52
Change from Baseline in Proteinuria Based on Spot Urine Protein-Creatinine Ratio | Baseline, Weeks 26, and 52
Change from Baseline in Proteinuria Based on Spot Urine Albumin-Creatinine Ratio | Baseline, Weeks 26, and 52
Change from Baseline in Hematuria | Baseline, Weeks 26, and 52

CONTACTS AND LOCATIONS:
Locations (66):
- Argentina (5):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, San Juan Bautista
  - Research Site, Santa Fe
- Australia (4):
  - Research Site, Clayton
  - Research Site, Heidelberg
  - Research Site, Nedlands
  - Research Site, Wollongong
- Brazil (5):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (6):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanchang
  - Research Site, Shenzhen
- France (4):
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Göttingen
  - Research Site, Ludwigshafen
  - Research Site, München
- Italy (4):
  - Research Site, Brescia
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Pisa
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Warsaw
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Pamplona
  - Research Site, San Sebastián de los Reyes
  - Research Site, Santander
  - Research Site, Seville
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (5):
  - Research Site, Altındağ
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Kocaeli
  - Research Site, Merkez
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR